CLINICAL TRIAL: NCT00793637
Title: Prospective Multicenter Case Series to Evaluate Handling and Possible Complications Related to the Angular Stable Locking System in Patients With Proximal and Distal Tibial, Femoral and Humeral Fractures Treated With Intramedullary Nails
Brief Title: Evaluation of Handling and Possible Complications Related to the Newly Developed Angular Stable Locking System (ASLS)
Acronym: ASLS-Pre
Status: Completed | Type: Observational
Sponsor: AO Clinical Investigation and Publishing Documentation (Other)
Collaborators: Synthes Inc. (Industry)
Responsible Party: Sponsor
Organization: AO Innovation Translation Center (Other)
Other Study IDs: ASLS-Pre-08
Record Dates: First submitted 2008-11-17; First posted 2008-11-19 (Estimated); Last update posted 2021-07-22 (Actual); Status verified 2009-08

CONDITIONS: Humerus Fracture; Femur Fracture; Tibia Fracture
Keywords: Angular stable locking system; Handling test; Complications
MeSH Terms: conditions — Humeral Fractures; Femoral Fractures; Tibial Fractures

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Surgical: Patients with proximal and/or distal tibial, femoral and/or humeral fractures treated with intramedullary nails and the Angular Stable Locking System(ASLS)

SUMMARY:
In many cases, the existing locking bolts and screws in intramedullary nails do not provide sufficient stability. Due to the play between screw and nail, the reduction can be lost and the instability can result in malunions, nonunions, or pseudoarthrosis. Consequently, secondary angular fracture dislocation (defined as a difference of the angle of 10° or more from the post-operative to the follow-up x-rays) can be observed in approximately 30% of patients after conventional intramedullary nailing of proximal third tibial fractures and in approximately 0-2% in patients with distal third tibial fractures. Therefore, an Angular Stable Locking System for Intramedullary Nails (ASLS) was developed to reduce the risk of secondary loss of reduction by providing axial and angular stability. ASLS provides angular stable fixation between nails and screws with resorbable sleeves used as dowels in the nail locking holes.

The present study evaluates the handling of ASLS and the surgeon's compliance as well as any complications occurring during the baseline and the follow-up period in patients with proximal and distal tibial, femoral and humeral fractures treated with intramedullary nails. Furthermore, the relationship of any occurred complications to ASLS will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* The patient is ≥ 18 years old
* One of the following bones is fractured so that the fracture is affecting the proximal or the distal third of the bone without affecting the joint surface: Humerus, Femur, Tibia
* The fracture is fixed with one of the following cannulated implants Humerus: Expert HN, Expert PHN. Femur: Expert LFN, Expert RAFN, CFN, DFN, AFN. Tibia: Expert TN, CTN.
* The patient is willing and able to participate in the study follow-up according to the CIP.
* The patient is able to understand and read local language at elementary level.
* The patient is willing and able to give written informed consent to participate in the study.

Exclusion criteria:

* The patient is legally incompetent.
* Preexistent malunion or nonunion of the bone that is planned to be treated with ASLS.
* The patient suffers from a polytrauma (multiple injuries, whereof one or the combination of several injuries is life-threatening).
* The patient suffers from active malignancy.
* The patient is affected by drug or alcohol abuse.
* The patient has participated in any other device or drug related clinical trial within the previous month.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: orthopedic clinics
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2008-08; Primary Completion 2009-07 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Surgeon's compliance and handling-oriented questionnaire | During surgery

SECONDARY OUTCOMES:
Rate of Complications | 6 months
General pain and pain at fracture site assessed by VAS | 6 months
Walking ability in patients with femoral or tibial fractures using the Parker mobility score | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Dankward Hoentzsch, MD, Principal Investigator — BG Unfallklinik Tübingen, 72076 Tübingen, Germany
Locations (4):
- Medizinische Universität Innsbruck, Abteilung Unfallchirurgie und Sporttraumatologie, Innsbruck, Austria
- Germany (3):
  - Charité - Universitätsmedizin Berlin, Centrum für Muskuloskeletale Chirurgie, Berlin
  - Universitätsklinikum Mainz, Klinik und Poliklinik für Unfallchirurgie, Mainz
  - BG Unfallklinik Tübingen, Tübingen